CLINICAL TRIAL: NCT04685031
Title: Ointment Therapy and Prevention of Cannulation-Induced Superficial Phlebitis
Acronym: OT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Komar University of Science and Technology (Other)
Responsible Party: Principal Investigator, yosra raziani, principal investigator,nursing department, Komar University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KomarUST
Record Dates: First submitted 2020-12-04; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Phlebitis
Keywords: Nitroglycerine; Clobetasol; phlebitis
MeSH Terms: conditions — Phlebitis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- nitroglycerin (Experimental): after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.
  Interventions: Drug: Nitroglycerin ointment; Drug: Clobetasol Topical
- clobetasol (Experimental): after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.
  Interventions: Drug: Nitroglycerin ointment; Drug: Clobetasol Topical
- routine (No Intervention): routine nursing care

INTERVENTIONS:
Drug: Nitroglycerin ointment — after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.
  Arms: clobetasol; nitroglycerin
Drug: Clobetasol Topical — after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.
  Arms: clobetasol; nitroglycerin

SUMMARY:
The aim of this study was to determine the effect of Clobetasol ointment with nitroglycerin ointment on the prevention of superficial phlebitis caused by cannulation. This clinical trial was conducted on 110 patients admitted to the surgical ward, in three groups of Clobetasol, nitroglycerin, and control. The data collection tools included demographic information, information about intravenous treatment and phlebitis measurement scale. In the intervention groups, after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.

DETAILED DESCRIPTION:
Aim: The aim of this study was to determine the effect of clobetasol ointment with nitroglycerin ointment on the prevention of superficial phlebitis caused by cannulation.

Background: Today, more than 80 to 90% of hospitalized patients receive intravenous treatment during their treatment, and more than 500 million peripheral venous catheters are placed annually, although cannulation provide numerous benefits in clinical setting, but because of its invasive feature, it can end in unpleasant outcomes such as phlebitis Method: This clinical trial was conducted on 110 patients admitted to the surgical ward, in three groups of clobetasol, nitroglycerin, and control. The data collection tools included demographic information, information about intravenous treatment and phlebitis measurement scale. In the intervention groups, after venipuncture, 1.5 cm (about 2 g) of ointment was applied in the distal part of the Angio catheter and the site was dressed with sterile gauze. In three time periods of 24, 48 and 72 hours from the time of venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* must be older than 18 years old
* must be in need of hospitalization at least 72 hours
* does not state any previous allergic reaction to the ointments
* does not use any types of drug that can hurts veins (chemotherapy drugs, diazepam. amiodarone, and....)

Exclusion Criteria:

* active infection
* discharge from hospital sooner than 72 hours
* displacement of cannula before 72 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Demographic information questionnaire | 72 hours
  age and type of disease

SECONDARY OUTCOMES:
The visual scale of phlebitis | 72hours
  The visual scale of phlebitis is as follows:
  Grade 0: no clinical symptoms, Grade 1: pain or redness, Grade 2: pain, redness or edema at the site, unclear vein boundaries, no rope vein in touch, Grade 3: pain, redness or edema at the site, clear blood vessels, no rope vein in touch, Grade 4: the presence of pain and erythema or edema at the site, the clearness of the arteries and the rope vein in touch.

IPD SHARING:
Plan to Share IPD: No